CLINICAL TRIAL: NCT06124404
Title: A Multicenter, Randomized, Single-blinded, Parallel, Two-step Trial to Evaluate the Effectiveness and Safety of Remimazolam Besylate for Injection for Sedation in ICU Patients
Brief Title: Step 1 of A Two-step Trial to Evaluate the Effectiveness and Safety of Remimazolam Besylate for Sedation in ICU Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Yichang Humanwell Pharmaceutical Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: WHUICU202205
Record Dates: First submitted 2023-09-29; First posted 2023-11-09 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-02

CONDITIONS: Mechanically Ventilated Patients

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Small dose (Experimental)
  Interventions: Drug: Remimazolam besylate
- Medium dose (Experimental)
  Interventions: Drug: Remimazolam besylate
- Large dose (Experimental)
  Interventions: Drug: Remimazolam besylate

INTERVENTIONS:
Drug: Remimazolam besylate — After a loading dose of 0.08mg/kg, a maintaining dose of 0.1mg/kg/h is given
  Other Names: A maintaining dose of 0.1mg/kg/h
  Arms: Small dose
Drug: Remimazolam besylate — After a loading dose of 0.08mg/kg, a maintaining dose of 0.2mg/kg/h is given
  Other Names: A maintaining dose of 0.2mg/kg/h
  Arms: Medium dose
Drug: Remimazolam besylate — After a loading dose of 0.08mg/kg, a maintaining dose of 0.4mg/kg/h is given
  Other Names: A maintaining dose of 0.4mg/kg/h
  Arms: Large dose

SUMMARY:
This is a Phase II, dose-escalation clinical trial conducted in mechanically ventilated patients receiving sedation no longer than 24 hours. The efficacy, safety, and pharmacokinetics of remimazolam besylate were evaluated using a randomized, single-blind design.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18 and ≤ 30 kg/m2
* Being Intubated and mechanically ventilated ≤48 hours before enrollment and expected to be on a ventilator for at least 6 hours
* Requirement for light to moderate sedation (a Richmond agitation-sedation scale score of -2 to 1)

Exclusion Criteria:

* Refusal to be included
* Allergy or unsuitability to any composition of study drugs or remifentanil
* Living expectancy less than 48 hours
* Myasthenia gravis
* Status asthmaticus
* Abdominal compartment syndrome
* Serious hepatic dysfunction (CTP 10-15);
* Chronic kidney disease with glomerular filtration rate (GFR) < 29 ml/min/1.73m2
* Mean blood pressure less than 65 mm Hg or the need for a continuous infusion of norepinephrine at ≥0.5 ug/kg/min to maintain Mean blood pressure ≥ 65 mm Hg
* Possible requirement for surgery or bedside tracheostomy in 24 hours
* Possible requirement for renal replacement therapy in 24 hours
* Acute severe neurological disorder and any other condition interfering with sedation assessment
* Abuse of controlled substances or alcohol
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The percentage of time in the target sedation range without rescue sedation | Within 24 hours while receiving the study drug
  The percentage of time in the target sedation range without rescue sedation

SECONDARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | Within 48 hours after the stop of the study drug
  The number and severity of treatment emergent adverse events (TEAEs)

OTHER OUTCOMES:
Cmax | Within 24 hours while receiving the study drug
  peak plasma concentration
The area under the plasma drug concentration-time curve | Within 24 hours while receiving the study drug
  The area under the plasma drug concentration-time curve (AUC)
t1/2 | Within 24 hours while receiving the study drug
  half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China